CLINICAL TRIAL: NCT04187950
Title: NECTAR Study: Nectar (Honey) Effects on Comfort, Thoughts, and Regularity
Acronym: NECTAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: National Honey Board (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 20121
Record Dates: First submitted 2019-10-02; First posted 2019-12-05 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Gastrointestinal Dysfunction; Physiological Stress; Cognition - Other
Keywords: gastrointestinal transit time, mood, emotion
MeSH Terms: interventions — Yogurt; Therapeutics

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, single-blind, crossover study with two 2-week treatment conditions separated by at least a 4-week washout period between conditions. Participant flow through the study conditions will be counterbalanced. Participants will be randomly allocated to yogurt with honey first or control first.
Who Masked: Participant
Masking Description: Participants will be blinded to the order in which they receive the study treatments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yogurt with inactivated B. lactis and added cane sugar (Placebo Comparator): Participants will consume yogurt with heat inactivated B. lactis and added cane sugar twice daily for 14 days.
  Interventions: Dietary Supplement: Yogurt with heat-inactivated B. lactis and added cane sugar
- Yogurt with B. lactis and added honey (Experimental): Participants will consume yogurt with B. lactis and added honey twice daily for 14 days.
  Interventions: Dietary Supplement: Yogurt with B. lactis and added honey

INTERVENTIONS:
Dietary Supplement: Yogurt with B. lactis and added honey — The intervention condition will utilize a commercially available yogurt (Activia) that contains Bifidobacterium animalis lactis DN-173 010/CNCM I-2494 (B. lactis). Participants will consume 170 g of yogurt with honey twice daily for 14 days.
  Other Names: Treatment
  Arms: Yogurt with B. lactis and added honey
Dietary Supplement: Yogurt with heat-inactivated B. lactis and added cane sugar — The control condition will utilize a commercially available yogurt (Activia) following heat inactivation of the probiotic Bifidobacterium animalis lactis DN-173 010/CNCM I-2494 (B. lactis). Participants will consume 170 g of the heat-inactivated yogurt with added cane sugar twice daily for 14 days.The added cane sugar will be an isocaloric amount to the honey.
  Other Names: Control
  Arms: Yogurt with inactivated B. lactis and added cane sugar

SUMMARY:
This study aims to test the central hypothesis that adding to the diet daily yogurt with honey provides beneficial effects on digestive health and subjective mood in healthy adults.

DETAILED DESCRIPTION:
This clinical trial will be a randomized, controlled, double-blind, crossover study with two 2-week treatment conditions separated by at least a 4-week washout period between conditions. Participant flow through the study conditions will be counterbalanced. Participants will be randomly allocated to yogurt with honey first or control first. Before beginning the first intervention period, participants will undergo a 2-week lead-in period that is devoid of all supplemental and dietary probiotics, fermented dairy products, and fermented foods. Participants will be asked to refrain from consuming all supplemental and dietary probiotics, fermented dairy products, and fermented foods throughout the entire study.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Between the ages of 22-64 years at the time of consent
* Body mass index of 18.5 to 29.9 kg/m^2.
* Normal or corrected-to-normal vision based on the minimal 20/20 standard in order to complete the cognitive task (below 20/20 vision).
* Ability to drop off fecal sample within 30 minutes of defecation
* Have between 3-6 bowel movements per week

Exclusion Criteria:

* Current pregnancy, lactation, or post-menopausal
* Tobacco use
* Honey allergy or intolerance
* Dairy allergy, lactose intolerance
* Food dye allergy/intolerance
* Prior physician diagnosed gastrointestinal disease (chronic constipation, diarrhea, Crohn's disease, celiac disease, ulcerative colitis, irritable bowel syndrome, diverticulosis, stomach or duodenal ulcers, hepatitis, or gastroesophageal reflux disease (GERD))
* Current use or use of antibiotics in the past 3 months
* Current use of any of the following types of medications: laxatives, anti-diarrhea medications, narcotics, enemas, antispasmodics, anticonvulsants, prescription proton pump inhibitors, prokinetic agents, histamine-2 Rc antagonists (prescription GERD medication)
* Body mass index > 29.9 kg/m^2
* Prior malabsorptive bariatric surgery (i.e. gastric bypass, sleeve gastrectomy)
* Restrictive bariatric surgery (i.e. adjustable gastric band) within the past 5 years
* Concurrent enrollment in another dietary, exercise, or medication study

Ages: 22 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2021-05-19 (Actual); Primary Completion 2022-11-02 (Actual); Study Completion 2022-11-02 (Actual)

PRIMARY OUTCOMES:
Intestinal transit time measured using colored dye markers | 2 weeks
  Determine the impact of consumption of daily yogurt with honey on intestinal transit time in vivo compared to control, yogurt containing heat-inactivated B.lactis with added sugar. Intestinal transit time will be measured using colored dye markers.

SECONDARY OUTCOMES:
Digestive health measured using daily stool records with the Bristol Stool Scale | 2 weeks
  Determine the impact of consumption of daily yogurt with honey on digestive health compared to control (yogurt containing heat-inactivated B. lactis) using daily stool records. Within the records, participants rate stool consistency using the Bristol Stool Scale.
Digestive health measured using rating scales of additional symptoms in daily stool records | 2 weeks
  Determine the impact of consumption of daily yogurt with honey on other measures of digestive health compared to control (yogurt containing heat-inactivated B. lactis) using daily stool records. Within the records, ratings of additional gastrointestinal symptoms include ease of passage, abdominal pain, bloating, burping, flatulence, nausea, reflux, and rumblings.
Digestive health measured using the Gastrointestinal Tolerability questionnaire | 2 weeks
  Determine the impact of consumption of daily yogurt with honey on other measures of digestive health compared to control (yogurt containing heat-inactivated B. lactis) using the Gastrointestinal Tolerability questionnaire. This questionnaire assesses gastrointestinal health through 6 questions related to gastrointestinal health including nausea, bloating, rumblings, gas/flatulence, abdominal pain, and diarrhea. Each of the questions pertains to experience of symptoms in the past 7 days.
Digestive health measured using the Gastrointestinal Quality of Life Index (GIQLI) questionnaire | 2 weeks
  Determine the impact of consumption of daily yogurt with honey on other measures of digestive health compared to control (yogurt containing heat-inactivated B. lactis) using the Gastrointestinal Quality of Life Index (GIQLI) questionnaire. The GIQLI assesses gastrointestinal health through a series of 36 questions pertaining to daily life and gastrointestinal symptoms experienced in the past 2 weeks.
Mood measured using the Emotional Image Task | 2 weeks
  Determine the impact of consumption of daily yogurt with honey on mood states compared to control (yogurt containing heat-inactivated B. lactis) using the Emotional Image Task. This task measures response to neutral, positive, and negative image stimuli using participant valence, arousal, and dominance ratings.
Mood measured using the Positive and Negative Affect Schedule (PANAS) questionnaire | 2 weeks
  Determine the impact of consumption of daily yogurt with honey on mood states compared to control (yogurt containing heat-inactivated B. lactis) using the Positive and Negative Affect Schedule (PANAS) questionnaire. The PANAS assesses general mood using a 20-item scale that includes words associated with either positive (10 words) or negative (10 words) emotions.
Mood measured using the Depression, Anxiety, and Stress Scales-42 (DASS-42) questionnaire | 2 weeks
  Determine the impact of consumption of daily yogurt with honey on mood states compared to control (yogurt containing heat-inactivated B. lactis) using the Depression, Anxiety, and Stress Scales-42 (DASS-42) questionnaire. The DASS-42 includes subscales with 42 questions regarding negative emotional states and is used to assess mental health over the past week.
Mood measured using Patient-Reported Outcomes Measurement Information System (PROMIS) questionnaires | 2 weeks
  Determine the impact of consumption of daily yogurt with honey on mood states compared to control (yogurt containing heat-inactivated B. lactis) using Patient-Reported Outcomes Measurement Information System (PROMIS) questionnaires. Specific PROMIS questionnaires utilized included PROMIS SF v1.0 - Anger 8a, PROMIS SF v1.0 - Anxiety 8a, PROMIS SF v1.0 - Fatigue 8a, PROMIS SF v1.0 - Positive Affect 15a, PROMIS SF v1.0 - Self-Efficacy Manage Emotions 8a, PROMIS SF v1.0 - Fatigue 13a (FACIT-Fatigue), PROMIS SF v1.1 - Global Health, and PROMIS SF v2.0 - Cognitive Function 8a. PROMIS. Surveys were scored using the recommended HealthMeasures Scoring Service.
Cognitive function assessed using the Spatial Reconstruction Task | 2 weeks
  Determine the impact of consumption of daily yogurt with honey on cognitive function compared to control (yogurt containing heat-inactivated B. lactis) using the Spatial Reconstruction Task. This task requires participants to successfully encode and retrieve information pertaining to the position of six objects in relation to each other, necessitating recruitment of the hippocampal memory system.
Gastrointestinal microbiota assessed using relative abundances | 2 weeks
  Determine the impact of daily consumption of yogurt with honey on the gastrointestinal microbiota compared to control (yogurt containing heat-inactivated B. lactis). Relative abundances of the gastrointestinal microbiota will be measured with 16S amplicon sequencing.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois at Urbana-Champaign, Urbana, Illinois, United States

REFERENCES:
- [Derived] Mysonhimer AR, Brown MD, Alvarado DA, Cornman E, Esmail M, Abdiel T, Gutierrez K, Vasquez J, Cannavale CN, Miller MJ, Khan NA, Holscher HD. Honey Added to Yogurt with Bifidobacterium animalis subsp. lactis DN-173 010/CNCM I-2494 Supports Probiotic Enrichment but Does Not Reduce Intestinal Transit Time in Healthy Adults: A Randomized, Controlled, Crossover Trial. J Nutr. 2024 Aug;154(8):2396-2410. doi: 10.1016/j.tjnut.2024.05.028. Epub 2024 Jun 1. PMID 38830472